CLINICAL TRIAL: NCT04776590
Title: Neoadjuvant Chemoradiotherapy Plus Tislelizumab Followed by Surgery for Thoracic Esophageal Squamous Cell Cancer: A Prospective, Single Arm, Pilot Study
Brief Title: Chemoradiotherapy Plus Immunotherapy Followed by Surgery for Esophageal Cancer
Acronym: CRISEC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, kunyu yang, Director of Department of Oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESC001
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Esophagus Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab arm (Experimental): Radiotherapy: PTV 41.4Gy in 23 Fractions，5 days per week; Chemotherapy: Paclitaxel (Albumin bound) (100mg per square meter of body-surface area weekly) and Caboplatin (area under the curve of 2 mg per milliliter per minute weekly) for 5 weeks, concurrent with radiotherapy; Immunotherapy: Tislelizumab (200mg per 3 weeks)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — neoadjuvant immunotherapy

SUMMARY:
Neoadjuvant chemoradiotherapy is recommended as standard therapy for resectable esophageal cancer. The recurrence rate after surgery following neoadjuvant chemoradiotherapy is about 35%. Whether achieving pathological complete response after neoadjuvant chemoradiotherapy is significantly associated with recurrence after surgery. It is reported that immunotherapy combined with chemotherapy improved survival compared with chemotherapy alone in first line therapy of advanced esophageal cancer. We hypothesize that the addition of immunotherapy to neoadjuvant chemoradiotherapy is helpful to improving pathologic complete response and survival.

ELIGIBILITY:
Main Inclusion Criteria:

* Pathologically diagnosed as esophageal squamous cell carcinoma
* Initially diagnosed as thoracic esophageal cancer
* resectable or potantially resectable
* II-IVA according to AJCC 8th edition；
* KPS≥70
* Adequate organ function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | 1 day on which pathologic results is reported
  Pathologic complete response rate

SECONDARY OUTCOMES:
Disease free survival | 2 years after surgery
  Disease free survival
overall survival | 2 years after enrollment
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kunyu Yang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zheng R, Zeng H, Zhang S, He J. Annual report on status of cancer in China, 2011. Chin J Cancer Res. 2015 Feb;27(1):2-12. doi: 10.3978/j.issn.1000-9604.2015.01.06. PMID 25717220
- [Background] Rice TW, Rusch VW, Apperson-Hansen C, Allen MS, Chen LQ, Hunter JG, Kesler KA, Law S, Lerut TE, Reed CE, Salo JA, Scott WJ, Swisher SG, Watson TJ, Blackstone EH. Worldwide esophageal cancer collaboration. Dis Esophagus. 2009;22(1):1-8. doi: 10.1111/j.1442-2050.2008.00901.x. PMID 19196264
- [Background] Rice TW, Chen LQ, Hofstetter WL, Smithers BM, Rusch VW, Wijnhoven BP, Chen KL, Davies AR, D'Journo XB, Kesler KA, Luketich JD, Ferguson MK, Rasanen JV, van Hillegersberg R, Fang W, Durand L, Cecconello I, Allum WH, Cerfolio RJ, Pera M, Griffin SM, Burger R, Liu JF, Allen MS, Law S, Watson TJ, Darling GE, Scott WJ, Duranceau A, Denlinger CE, Schipper PH, Lerut TE, Orringer MB, Ishwaran H, Apperson-Hansen C, DiPaola LM, Semple ME, Blackstone EH. Worldwide Esophageal Cancer Collaboration: pathologic staging data. Dis Esophagus. 2016 Oct;29(7):724-733. doi: 10.1111/dote.12520. PMID 27731547
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Mariette C, Balon JM, Piessen G, Fabre S, Van Seuningen I, Triboulet JP. Pattern of recurrence following complete resection of esophageal carcinoma and factors predictive of recurrent disease. Cancer. 2003 Apr 1;97(7):1616-23. doi: 10.1002/cncr.11228. PMID 12655517
- [Background] Dresner SM, Griffin SM. Pattern of recurrence following radical oesophagectomy with two-field lymphadenectomy. Br J Surg. 2000 Oct;87(10):1426-33. doi: 10.1046/j.1365-2168.2000.01541.x. PMID 11044172
- [Background] Liu Q, Cai XW, Wu B, Zhu ZF, Chen HQ, Fu XL. Patterns of failure after radical surgery among patients with thoracic esophageal squamous cell carcinoma: implications for the clinical target volume design of postoperative radiotherapy. PLoS One. 2014 May 12;9(5):e97225. doi: 10.1371/journal.pone.0097225. eCollection 2014. PMID 24820177
- [Background] Oppedijk V, van der Gaast A, van Lanschot JJ, van Hagen P, van Os R, van Rij CM, van der Sangen MJ, Beukema JC, Rutten H, Spruit PH, Reinders JG, Richel DJ, van Berge Henegouwen MI, Hulshof MC. Patterns of recurrence after surgery alone versus preoperative chemoradiotherapy and surgery in the CROSS trials. J Clin Oncol. 2014 Feb 10;32(5):385-91. doi: 10.1200/JCO.2013.51.2186. Epub 2014 Jan 13. PMID 24419108
- [Background] Law S, Fok M, Chow S, Chu KM, Wong J. Preoperative chemotherapy versus surgical therapy alone for squamous cell carcinoma of the esophagus: a prospective randomized trial. J Thorac Cardiovasc Surg. 1997 Aug;114(2):210-7. doi: 10.1016/S0022-5223(97)70147-8. PMID 9270638
- [Background] Ancona E, Ruol A, Santi S, Merigliano S, Sileni VC, Koussis H, Zaninotto G, Bonavina L, Peracchia A. Only pathologic complete response to neoadjuvant chemotherapy improves significantly the long term survival of patients with resectable esophageal squamous cell carcinoma: final report of a randomized, controlled trial of preoperative chemotherapy versus surgery alone. Cancer. 2001 Jun 1;91(11):2165-74. PMID 11391598
- [Background] Allum WH, Stenning SP, Bancewicz J, Clark PI, Langley RE. Long-term results of a randomized trial of surgery with or without preoperative chemotherapy in esophageal cancer. J Clin Oncol. 2009 Oct 20;27(30):5062-7. doi: 10.1200/JCO.2009.22.2083. Epub 2009 Sep 21. PMID 19770374
- [Background] Kelsen DP, Winter KA, Gunderson LL, Mortimer J, Estes NC, Haller DG, Ajani JA, Kocha W, Minsky BD, Roth JA, Willett CG; Radiation Therapy Oncology Group; USA Intergroup. Long-term results of RTOG trial 8911 (USA Intergroup 113): a random assignment trial comparison of chemotherapy followed by surgery compared with surgery alone for esophageal cancer. J Clin Oncol. 2007 Aug 20;25(24):3719-25. doi: 10.1200/JCO.2006.10.4760. PMID 17704421
- [Background] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Background] Boonstra JJ, Kok TC, Wijnhoven BP, van Heijl M, van Berge Henegouwen MI, Ten Kate FJ, Siersema PD, Dinjens WN, van Lanschot JJ, Tilanus HW, van der Gaast A. Chemotherapy followed by surgery versus surgery alone in patients with resectable oesophageal squamous cell carcinoma: long-term results of a randomized controlled trial. BMC Cancer. 2011 May 19;11:181. doi: 10.1186/1471-2407-11-181. PMID 21595951
- [Background] Gebski V, Burmeister B, Smithers BM, Foo K, Zalcberg J, Simes J; Australasian Gastro-Intestinal Trials Group. Survival benefits from neoadjuvant chemoradiotherapy or chemotherapy in oesophageal carcinoma: a meta-analysis. Lancet Oncol. 2007 Mar;8(3):226-34. doi: 10.1016/S1470-2045(07)70039-6. PMID 17329193
- [Background] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Donahue JM, Nichols FC, Li Z, Schomas DA, Allen MS, Cassivi SD, Jatoi A, Miller RC, Wigle DA, Shen KR, Deschamps C. Complete pathologic response after neoadjuvant chemoradiotherapy for esophageal cancer is associated with enhanced survival. Ann Thorac Surg. 2009 Feb;87(2):392-8; discussion 398-9. doi: 10.1016/j.athoracsur.2008.11.001. PMID 19161745
- [Background] Schneider PM, Baldus SE, Metzger R, Kocher M, Bongartz R, Bollschweiler E, Schaefer H, Thiele J, Dienes HP, Mueller RP, Hoelscher AH. Histomorphologic tumor regression and lymph node metastases determine prognosis following neoadjuvant radiochemotherapy for esophageal cancer: implications for response classification. Ann Surg. 2005 Nov;242(5):684-92. doi: 10.1097/01.sla.0000186170.38348.7b. PMID 16244542
- [Background] Leng X, He W, Yang H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Liu H, Yang H, Li T, Zhang X, Li Q, Wang G, Mao T, Guo X, Lin T, Liu M, Fu J, Han Y. Prognostic Impact of Postoperative Lymph Node Metastases After Neoadjuvant Chemoradiotherapy for Locally Advanced Squamous Cell Carcinoma of Esophagus: From the Results of NEOCRTEC5010, a Randomized Multicenter Study. Ann Surg. 2021 Dec 1;274(6):e1022-e1029. doi: 10.1097/SLA.0000000000003727. PMID 31855875
- [Derived] Yang J, Huang A, Yang K, Jiang K. Neoadjuvant chemoradiotherapy plus tislelizumab followed by surgery for esophageal carcinoma (CRISEC study): the protocol of a prospective, single-arm, phase II trial. BMC Cancer. 2023 Mar 15;23(1):249. doi: 10.1186/s12885-023-10687-8. PMID 36922805